CLINICAL TRIAL: NCT05633134
Title: Precision Preoperative Embolization of Pelvic Tumors to Improve Surgical Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhi Xin, Doctor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPE-PT
Record Dates: First submitted 2022-11-20; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Embolization; Pelvic Tumor
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision preoperative embolization (Experimental): 60 patients with pelvic tumors will undergo arteriography and receive transcatheter arterial embolization of pelvic tumors 0-24 hours prior to surgery.
  Interventions: Procedure: Arteriography and precision preoperative embolization
- Control group (Active Comparator): 60 patients with pelvic tumors will undergo arteriography and without transcatheter arterial embolization of pelvic tumors prior to surgery.
  Interventions: Procedure: Arteriography

INTERVENTIONS:
Procedure: Arteriography and precision preoperative embolization — Arteriography and transcatheter arterial embolization of pelvic tumors 0-24 hours prior to surgery.
  Other Names: Transcatheter arterial embolization; Therapeutic angiography; Selective arterial embolization
  Arms: Precision preoperative embolization
Procedure: Arteriography — Arteriography of pelvic tumors 0-24 hours prior to surgery.
  Arms: Control group

SUMMARY:
The main purpose of this study is to assess the efficacy of precision preoperative embolization in decreasing operative blood loss, reducing surgical complications in pelvic tumor surgery. Furthermore the study aims at describing the vascularity in a series of pelvic tumors, and to correlate this with perioperative blood loss.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of precision preoperative embolization in decreasing operative blood loss, reducing surgical complications in pelvic tumor surgery，which including poor wound healing，nerve injury，and pelvic organs dysfunction. Furthermore the study aims at describing the vascularity in a series of pelvic tumors,which contains four grade：poor，moderate，rich and abundant and to correlate this with perioperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic pelvic tumor
* Confirmed by contrast-enhanced magnetic resonance imaging (MRI) or computed tomography (CT) of the pelvic
* Planned surgical resection

Exclusion Criteria:

* Contrast medium allergy
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood loss | Measured intraoperatively
  Perioperative blood loss measured intraoperatively

SECONDARY OUTCOMES:
Adverse events related to angiography or embolization | Within 2 postoperative days
  Including symptoms of nerve compression, pelvic organ ischemia injury
Adverse events related to surgery | Within 30 postoperative days
  including poor wound healing，nerve injury，pelvic organ dysfunction
Vascularization grade of pelvic tumors | At the angiographic procedure prior to embolization performed 0-24 hours before surgery
  it contains four grades：poor、moderate、rich、abundant
postoperative blood loss | Within 2 postoperative days
  blood loss measured through the drainage within 2 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: XIN ZHI, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No